CLINICAL TRIAL: NCT03791840
Title: The Accuracy of High-resolution Ultrasound in the Detection of Lymph Node Metastasis From Breast Cancer and the Proposal of Node Imaging Reporting and Data System
Brief Title: The Value of High-resolution Ultrasound in the Detection of Lymph Node Metastasis: a Proposal of NI-RADS
Acronym: NI-RADS
Status: Completed | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, HP Yang, Clinical Professor, Peking University People's Hospital
Other Study IDs: PKUPHUS002
Record Dates: First submitted 2018-12-31; First posted 2019-01-03 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Breast Neoplasms
Keywords: breast neoplasms; Ultrasonography, Interventional; Biopsy, Large-Core Needle; Biopsy, Fine-Needle
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Fresh lymph node specimens from breast cancer patients were detected using ultrasound.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Ultrasound evaluation: Eligible patients undergo lymph node biopsy or lymph node dissection. Before surgery, the status of axillary lymph node status was evaluated using ultrasound. After surgery, all lymph node specimens would be collected and be assessed using ultrasound in a special evaluation system in vitro.
  Interventions: Diagnostic Test: Ultrasound evaluation

INTERVENTIONS:
Diagnostic Test: Ultrasound evaluation — High-frequency ultrasound is used to detected the lymph node metastasis in vivo and vitro. The lymph node number, morphology and elastographic parameters are collected in the patients and in fresh lymph node specimens.

SUMMARY:
The status of axillary lymph node (ALN) is an important reference indicator for breast cancer surgery and systemic treatment, which is also an important prognostic indicator for breast cancer. Therefore, it is extremely important for surgeons to accurately determine whether axillary lymph nodes have metastasis and the number of metastatic lymph nodes. The value of ultrasound diagnosing the status of axillary lymph nodes was controversial in recent publications. Therefore, there is a high need to prove the accuracy and precision of ultrasound for axillary lymph node metastasis in breast cancer patients. The aim of this study is to assess the usefulness of ultrasound in the diagnosis of axillary lymph node status in breast cancer patients by gathering in vivo and vitro ultrasonographic parameters to build a clinical useful categorization system

DETAILED DESCRIPTION:
To facilitate the non-invasive assessment of lymph node status preoperatively, we use ultrasound to detect lymph node metastasis. We designed this study to obtain in vivo and vitro ultrasound features and parameters. Before surgery, the detailed ultrasound features are collected during routine ultrasound examination. After the completion of the axillary surgery, fresh lymph node specimens are collected for in vitro ultrasound evaluation one by one in a specially-designed detection system. Statistical models are built to categorize the probability of metastasis of lymph node according to a proposed categorization system similar as BI-RADS(Breast Imaging Reporting and Data System), which is named NI-RADS (Node Imaging Reporting and Data System).

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer.
* Pathological axillary lymph node staging planned.
* Axillary lymph node not removed prior to the study.

Exclusion Criteria:

* Refusal participation in the study.

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with invasive breast cancer planned to receive surgical axillary lymph node staging are eligible.
Sampling Method: Probability Sample
Enrollment: 135 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Sensitivity of ultrasound | Through study completion, an average of 1 year.
  True positive rate measures the proportion of positives that are correctly identified by ultrasound

SECONDARY OUTCOMES:
Specificity of ultrasound | Through study completion, an average of 1 year.
  The true negative rate measures the proportion of negatives that are correctly identified.
Diagnostic model of lymph node ultrasound | Through study completion, an average of 1 year
  A diagnostic model or nomogram would be developed to facilitate the diagnosis of the lymph node ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Shu Wang, MD, Principal Investigator — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Han P, Yang H, Liu M, Cheng L, Wang S, Tong F, Liu P, Zhou B, Cao Y, Liu H, Wang C, Peng Y, Shen D, Wang S. Lymph Node Predictive Model with in Vitro Ultrasound Features for Breast Cancer Lymph Node Metastasis. Ultrasound Med Biol. 2020 Jun;46(6):1395-1402. doi: 10.1016/j.ultrasmedbio.2020.01.030. Epub 2020 Mar 5. PMID 32146007